CLINICAL TRIAL: NCT02690610
Title: Value of Rapid on Site Evaluation During Endobronchial Ultrasound Guided Trans-bronchial Needle Aspiration (EBUS-TBNA) in the Diagnosis of Mediastinal Lesions
Brief Title: Value of Rapid on Site Evaluation During EBUS-guided TBNA in the Diagnosis of Mediastinal Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Adel Salah Bediwy, Professor, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 30613/11/15
Record Dates: First submitted 2016-01-30; First posted 2016-02-24 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Mediastinum
Keywords: EBUS, Mediastinal lesions, Mediastinal lymph node

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with mediastinal lesions (Experimental): EBUS TBNA of mediastinal lesions or lymph nodes
  Interventions: Procedure: EBUS TBNA of mediastinal lesions or lymph nodes

INTERVENTIONS:
Procedure: EBUS TBNA of mediastinal lesions or lymph nodes — Through endo-bronchial ultrasound, a transbronchial needle will be introduced to take biopsies from mediastinal lesions under ultrasonic guidance.

SUMMARY:
This prospective study will include 30 patients with hilar/mediastinal lymph nodes detected by thoracic CT either there was a known lung malignancy (for staging purpose) or not (for diagnosing purpose).

All patients will undergo to ROSE during EBUS-guided TBNA. Mediastinoscopy or other invasive procedures will be performed if EBUS-guided TBNA doesn't provide representative material.

DETAILED DESCRIPTION:
All patients will be subjected to the following parameters:

1. Thorough history taking and full clinical examination.
2. Chest X-ray (postro-anterior and lateral views) before and after the procedure.
3. Recent Computed Tomography (CT chest) with contrast.
4. Laboratory studies:

   * Complete liver functions.
   * Blood urea and serum creatinine.
   * Complete blood picture (including platelet count).
   * Erythrocyte sedimentation rate (ESR).
   * Fasting and postprandial blood sugar.
5. Preoperative evaluation: Pulmonary function tests (PFT), Electrocardiogram (ECG), arterial blood gases (ABG) and coagulation profile (including bleeding & clotting times, prothrombin time& activity and activated partial thromboplastin time (APTT)) and oral anticoagulants should be stopped before the procedure for at least 48 hours.
6. Color doppler ultrasound in suspected vascular lesions.
7. Clinical and radiological follow up of patients over 1 week after the procedure to detect the occurrence of any complications.
8. The biopsy samples will be examined histopathologically. EBUS-TBNA will be done within 10 days of CT examination under local anesthesia and conscious sedation.

Convex Probe EBUS- Guided TBNA EBUS-guided TBNA examinations will be performed at both Tanta University Educational Hospital and Kobry Elkoba Military Hospital using Pantex EBUS probe and Hitachi ultrasound in the supine position under local anesthesia with lidocaine and conscious sedation.

Lymph nodes will be identified according to the Mountain's regional lymph node classification system (17). The lymph node stations of 2, 4, 7, 10 and 11 were evaluated systematically. During the process for every detected lymph node; short and long axis diameters, station of the lymph node, number of passes per patient and per lymph node were recorded for each patient.

N3 nodes will be sampled first and then N2 nodes to avoid contamination in lung cancer patients. The materials obtained by EBUS-guided TBNA will be smeared on slides. These slides will be air-dried and Diff-Quik (American Scientific Products, McGaw Park, IL) staining will be used for ROSE. Additional smears will be prepared for Papanicolaou staining and any remaining sample will be placed in 10% formalin for histologic evaluation. The results of ROSE were compared with the results of the final pathologic diagnosis. (17) Aspiration specimen was considered "insufficient" if there were not an adequate number of lymphocytes on the smear. Diagnosis as "malignant" in cytologic examination was considered as the "final diagnosis". For the patients whose EBUS-guided TBNA results were negative for malignancy, more invasive procedures such as mediastinoscopy will be done to confirm the diagnosis or radiologic follow-up on the outcome of the LNs for at least 6 months. On follow-up, LNs that persisted in size, diminished, or resolved were considered benign. A diagnosis of tuberculosis or sarcoidosis will be made based on cytopathology that showed the presence of caseating or noncaseating granuloma, in addition to clinical, radiological, and microbiological findings.

Any unexpected risk will be cleared to the participant and to Ethics committee. Waste materials will be disposed properly. All patients will sign an informed written consent. Patients' names will not be used and will be replaced by code numbers to confirm their privacy. Also, the results of the study will be used only for scientific purpose.

ELIGIBILITY:
Inclusion Criteria:

* Hilar/mediastinal lymph nodes with a short axis more than 1 cm on thoracic CT scan and/or PET-CT suspicious for malignancy with or without known lung malignancy.
* Hilar and/or mediastinal lymph nodes positive on PET/CT scan without regarding the diameter suspicious for malignancy.
* Recurrence or restaging of NSCLC after chemotherapy or radiation.
* Diagnosis of lung cancer when there is no endobronchial lesion.
* Diagnosis of both benign (especially tuberculosis and sarcoidosis) and malignant mediastinal lesions (eg. thymoma).

Exclusion Criteria:

* Cardiovascular instability.
* Lack of patient cooperation, e.g. intractable cough, inability to remain motionless or altered consciousness.
* Bleeding diathesis (activated partial thromboplastin time (APTT) ratio or international normalized ratio (INR) <1.3 or platelet count of <50000 per mm3).
* Respiratory failure and patient on mechanical ventilation.
* Severe chronic obstructive pulmonary disease (COPD) (FEV1<1 liter or <35% predicted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with accurate diagnosis of mediastinal lesions in relation to the total number studied. | 4-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Adel Salah Bediwy, MD, Study Chair — Chest Department, Faculty of Medicine, Tanta University
Locations (1):
- Chest Department, Faculty of Medicine, Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Herth FJ, Rabe KF, Gasparini S, Annema JT. Transbronchial and transoesophageal (ultrasound-guided) needle aspirations for the analysis of mediastinal lesions. Eur Respir J. 2006 Dec;28(6):1264-75. doi: 10.1183/09031936.00013806. PMID 17138681
- [Result] Herth FJ, Krasnik M, Kahn N, Eberhardt R, Ernst A. Combined endoscopic-endobronchial ultrasound-guided fine-needle aspiration of mediastinal lymph nodes through a single bronchoscope in 150 patients with suspected lung cancer. Chest. 2010 Oct;138(4):790-4. doi: 10.1378/chest.09-2149. Epub 2010 Feb 12. PMID 20154073
- [Result] Geake J, Hammerschlag G, Nguyen P, Wallbridge P, Jenkin GA, Korman TM, Jennings B, Johnson DF, Irving LB, Farmer M, Steinfort DP. Utility of EBUS-TBNA for diagnosis of mediastinal tuberculous lymphadenitis: a multicentre Australian experience. J Thorac Dis. 2015 Mar;7(3):439-48. doi: 10.3978/j.issn.2072-1439.2015.01.33. PMID 25922723
- [Result] Cardoso AV, Neves I, Magalhaes A, Sucena M, Barroca H, Fernandes G. The value of rapid on-site evaluation during EBUS-TBNA. Rev Port Pneumol (2006). 2015 Sep-Oct;21(5):253-8. doi: 10.1016/j.rppnen.2015.02.003. Epub 2015 Apr 1. PMID 25926258